CLINICAL TRIAL: NCT02478476
Title: DNA Single Nucleotide Polymorphisms as Predictors of Platinum and Taxane Related Adverse Events in Ovarian, Fallopian Tube, and Peritoneal Cancer Patients
Brief Title: DNA Single Nucleotide Polymorphisms as Predictors of Toxicity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: OvaGene Oncology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRBNet#673096
Record Dates: First submitted 2015-06-16; First posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The presence of single nucleotide polymorphisms (SNPs) in genes involved in platinum and taxane metabolism and detoxification have been correlated to increased risk of severe adverse events (AEs) when patients receive these drugs. The investigators propose studies to validate a comprehensive panel of twelve SNPs in ovarian cancer patients that may predict AEs when treated with therapies that include platinum and taxanes. Using these results to stratify patients to different dosing regimens, routes of administration, or in recurrent cancer to aid in drug selection, may improve outcome and reduce costs for the management of drug related side effects while not changing standard of care. Since these differences can be detected from blood, the determination of genotypes can be done using a standard blood sample taken after ovarian cancer is confirmed on the patient's pathology report. These genetic differences can be detected by QPCR and Next Generation Sequencing.

DETAILED DESCRIPTION:
The majority of ovarian cancer patients are treated with a combination of platinum- and taxane-based chemotherapy. While initial response rates are high (>90%), some patients experience severe AEs which can lead to discontinuation of therapy. However, both GOG and the paclitaxel package insert include treatment guidelines that involve a decreased dose regimen if AEs are encountered [1, 2]. The clinical validation of the genetic differences in these genes as biomarkers for severe AEs would allow the treating physician to alter dosing, thus increasing the time a patient could remain on the drug while decreasing side effects and unnecessary morbidity.

Another clinical utility of these genetic differences in ovarian cancer patient care is in the identification of which patients may not benefit from intraperitoneal (IP) chemotherapy or dose dense chemotherapy. While IP chemotherapy has been shown to improve patient outcome, the side effects are much more frequent and severe due to the high dose [3]. Testing the patients prior to treatment for predictive genotypes may factor into a doctor's decision to forego IP chemotherapy in favor of standard intravenous delivery. Dose dense chemotherapy has demonstrated improvements in outcome but also some increases in side effects [4, 5]. In both therapy regimens, the ability to stratify patients based on the risks of toxicities associated with treatment may lead to a greater benefit of IP or dose dense therapy while minimizing side effects and associated health care costs.

Previous studies in ovarian cancer have demonstrated that expression of the proteins ERCC1, GST, and p53 can affect the response to platinum based therapies in ovarian cancer patients [6-13]. When SNPs in the genes that encode these proteins were evaluated, a correlation to AEs in response to platinum-based therapies was made [14, 15]. Mutations that affected activity of ERCC1 were associated with nephrotoxicity. Mutations in GST family members were associated with neutropenia (GSTA1), neuropathy (GSTM3 and GSTP1), or anemia and thrombocytopenia (GSTM3). Mutations in p53 were associated with neutropenia. In these studies, mutations in XPD and XRCC1 were also found to be predictive of neutropenia (both XPD and XRCC1) and anemia (XPD only). More recently, a study done by the Scottish Gynecological Clinical Trials Group identified SNPs in BCL2, Current Version Date: 04/01/15 Previous Version Date: N/A, Initial version Page 6 of 23 OPRM1 SOX10 and TRPV1 that were associated with neurotoxicity [16]. Both the individual and combined value of these biomarkers needs to be assessed.

Reviewing studies done in other tumor types has identified SNPs associated with toxicities that may also be applicable in ovarian cancer. In breast cancer, SNPs in the CYP2C8, CYP17A1, and ABCG1 genes have been associated with an increased risk of grade 2+ peripheral neuropathy in patients treated with taxane-based therapies. [17, 18]. A different SNP in CYP17A1 (rs619824) has also been previously reported to be associated with bortezomib-induced neuropathy in multiple myeloma patients, potentially supporting the role of this protein in the onset of neuropathy [19]. Since these SNPs are germ line differences, there is reason to believe they may be valuable biomarkers in ovarian cancer also. In multiple myeloma, it has been suggested that identification and closer monitoring of patients at risk for neuropathy could be beneficial [20]. A similar strategy could be used with ovarian cancer patients to reduce severe toxicities that results in discontinuation of an effective drug.

The detection of these polymorphisms by QPCR has been confirmed by direct sequencing of cell lines and tumor tissue. The protocol has been tested in our research lab and has been validated in our CLIA regulated lab for both formalin fixed paraffin embedded samples and blood. In brief, DNA is purified over a spin column, quantitated, and mixed with a specific SNP assay and Master Mix (Life Technologies). Results were analyzed in the Life Technologies TaqMan Genotyper software version 1.3 to determine genotype. The SNPs were detected in blood samples collected from ovarian cancer patients and FFPE ovarian cancer specimens with similar frequencies as reported in the papers referenced above. SNPs from other tumor types were detected in the same blood samples from ovarian cancer patients or FFPE ovarian cancer specimens as well as in blood and FFPE samples from endometrial cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Female, greater than or equal to 18 years of age.
2. Must have pathologically confirmed ovarian, fallopian tube, or primary peritoneal cancer.
3. Able to provide a blood sample (3-5ml).
4. Planned course of therapy includes a platinum and/or taxane based chemotherapy.

Exclusion Criteria:

1. Has a clinically significant (per judgment of the PI) neurodegenerative, hematological, or cardiac related disease.
2. Has received prior chemotherapy.
3. Unable or unwilling to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pathologically confirmed ovarian, fallopian tube, or peritoneal cancer scheduled to receive platinum and/or taxane based chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of chemotherapy related toxicities including Anemia, Nephrotoxicity, Neutropenia, Neuropathy, and Thrombocytopenia associated with genotype. | one year
  Specific genotypes will be evaluated as predictors of toxicity when patients receive platinum and/or taxane based chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: William Ricketts, PhD, Study Director — OvaGene Oncology
Locations (1):
- Florida Hospital Cancer Institute, Orlando, Florida, United States

REFERENCES:
- [Background] Paclitaxel, [package insert], Bristol-Meyers Squibb Company, Princeton, NJ, April 2011.
- [Background] Chemotherapy procedure Manual, Gynecologic Oncology Group, January 2004.
- [Background] Wenzel LB, Huang HQ, Armstrong DK, Walker JL, Cella D; Gynecologic Oncology Group. Health-related quality of life during and after intraperitoneal versus intravenous chemotherapy for optimally debulked ovarian cancer: a Gynecologic Oncology Group Study. J Clin Oncol. 2007 Feb 1;25(4):437-43. doi: 10.1200/JCO.2006.07.3494. PMID 17264340
- [Background] Katsumata N, Yasuda M, Takahashi F, Isonishi S, Jobo T, Aoki D, Tsuda H, Sugiyama T, Kodama S, Kimura E, Ochiai K, Noda K; Japanese Gynecologic Oncology Group. Dose-dense paclitaxel once a week in combination with carboplatin every 3 weeks for advanced ovarian cancer: a phase 3, open-label, randomised controlled trial. Lancet. 2009 Oct 17;374(9698):1331-8. doi: 10.1016/S0140-6736(09)61157-0. Epub 2009 Sep 18. PMID 19767092
- [Background] Glaze S, Teitelbaum L, Chu P, Ghatage P, Nation J, Nelson G. Dose-dense paclitaxel with carboplatin for advanced ovarian cancer: a feasible treatment alternative. J Obstet Gynaecol Can. 2013 Jan;35(1):61-7. doi: 10.1016/s1701-2163(15)31050-1. PMID 23343799
- [Background] Milovic-Kovacevic M, Srdic-Rajic T, Radulovic S, Bjelogrlic S, Gavrilovic D. Expression of ERCC1 protein in biopsy specimen predicts survival in advanced ovarian cancer patients treated with platinum-based chemotherapy. J BUON. 2011 Oct-Dec;16(4):708-14. PMID 22331726
- [Background] Scheil-Bertram S, Tylus-Schaaf P, du Bois A, Harter P, Oppitz M, Ewald-Riegler N, Fisseler-Eckhoff A. Excision repair cross-complementation group 1 protein overexpression as a predictor of poor survival for high-grade serous ovarian adenocarcinoma. Gynecol Oncol. 2010 Nov;119(2):325-31. doi: 10.1016/j.ygyno.2010.07.018. Epub 2010 Aug 21. PMID 20728204
- [Background] Steffensen KD, Waldstrom M, Jakobsen A. The relationship of platinum resistance and ERCC1 protein expression in epithelial ovarian cancer. Int J Gynecol Cancer. 2009 Jul;19(5):820-5. doi: 10.1111/IGC.0b013e3181a12e09. PMID 19574766
- [Background] Steffensen KD, Waldstrom M, Jeppesen U, Brandslund I, Jakobsen A. Prediction of response to chemotherapy by ERCC1 immunohistochemistry and ERCC1 polymorphism in ovarian cancer. Int J Gynecol Cancer. 2008 Jul-Aug;18(4):702-10. doi: 10.1111/j.1525-1438.2007.01068.x. Epub 2007 Oct 24. PMID 17961161
- [Background] Hirazono K, Shinozuka T, Kuroshima Y, Itoh H, Kawai K. Immunohistochemical expression of glutathione S-transferase pi (GST-pi) and chemotherapy response in malignant ovarian tumors. J Obstet Gynaecol (Tokyo 1995). 1995 Jun;21(3):305-12. doi: 10.1111/j.1447-0756.1995.tb01015.x. PMID 8590371
- [Background] Howells RE, Dhar KK, Hoban PR, Jones PW, Fryer AA, Redman CW, Strange RC. Association between glutathione-S-transferase GSTP1 genotypes, GSTP1 over-expression, and outcome in epithelial ovarian cancer. Int J Gynecol Cancer. 2004 Mar-Apr;14(2):242-50. doi: 10.1111/j.1048-891X.2004.014207.x. PMID 15086723
- [Background] Bali A, O'Brien PM, Edwards LS, Sutherland RL, Hacker NF, Henshall SM. Cyclin D1, p53, and p21Waf1/Cip1 expression is predictive of poor clinical outcome in serous epithelial ovarian cancer. Clin Cancer Res. 2004 Aug 1;10(15):5168-77. doi: 10.1158/1078-0432.CCR-03-0751. PMID 15297421
- [Background] Ferrandina G, Fagotti A, Salerno MG, Natali PG, Mottolese M, Maneschi F, De Pasqua A, Benedetti-Panici P, Mancuso S, Scambia G. p53 overexpression is associated with cytoreduction and response to chemotherapy in ovarian cancer. Br J Cancer. 1999 Oct;81(4):733-40. doi: 10.1038/sj.bjc.6690756. PMID 10574264
- [Background] Khrunin AV, Moisseev A, Gorbunova V, Limborska S. Genetic polymorphisms and the efficacy and toxicity of cisplatin-based chemotherapy in ovarian cancer patients. Pharmacogenomics J. 2010 Feb;10(1):54-61. doi: 10.1038/tpj.2009.45. Epub 2009 Sep 29. PMID 19786980
- [Background] Sakano S, Hinoda Y, Sasaki M, Wada T, Matsumoto H, Eguchi S, Shinohara A, Kawai Y, Hara T, Nagao K, Hara T, Naito K, Matsuyama H. Nucleotide excision repair gene polymorphisms may predict acute toxicity in patients treated with chemoradiotherapy for bladder cancer. Pharmacogenomics. 2010 Oct;11(10):1377-87. doi: 10.2217/pgs.10.106. PMID 21047201
- [Background] McWhinney-Glass S, Winham SJ, Hertz DL, Yen Revollo J, Paul J, He Y, Brown R, Motsinger-Reif AA, McLeod HL; Scottish Gynaecological Clinical Trials Group. Cumulative genetic risk predicts platinum/taxane-induced neurotoxicity. Clin Cancer Res. 2013 Oct 15;19(20):5769-76. doi: 10.1158/1078-0432.CCR-13-0774. Epub 2013 Aug 20. PMID 23963862
- [Background] Hertz DL, Motsinger-Reif AA, Drobish A, Winham SJ, McLeod HL, Carey LA, Dees EC. CYP2C8*3 predicts benefit/risk profile in breast cancer patients receiving neoadjuvant paclitaxel. Breast Cancer Res Treat. 2012 Jul;134(1):401-10. doi: 10.1007/s10549-012-2054-0. Epub 2012 Apr 18. PMID 22527101
- [Background] Hertz DL, Roy S, Motsinger-Reif AA, Drobish A, Clark LS, McLeod HL, Carey LA, Dees EC. CYP2C8*3 increases risk of neuropathy in breast cancer patients treated with paclitaxel. Ann Oncol. 2013 Jun;24(6):1472-8. doi: 10.1093/annonc/mdt018. Epub 2013 Feb 14. PMID 23413280
- [Background] Corthals SL, Kuiper R, Johnson DC, Sonneveld P, Hajek R, van der Holt B, Magrangeas F, Goldschmidt H, Morgan GJ, Avet-Loiseau H. Genetic factors underlying the risk of bortezomib induced peripheral neuropathy in multiple myeloma patients. Haematologica. 2011 Nov;96(11):1728-32. doi: 10.3324/haematol.2011.041434. Epub 2011 Jul 26. PMID 21791469
- [Background] Velasco R, Petit J, Clapes V, Verdu E, Navarro X, Bruna J. Neurological monitoring reduces the incidence of bortezomib-induced peripheral neuropathy in multiple myeloma patients. J Peripher Nerv Syst. 2010 Mar;15(1):17-25. doi: 10.1111/j.1529-8027.2010.00248.x. PMID 20433602
- [Background] Pike CT, Birnbaum HG, Muehlenbein CE, Pohl GM, Natale RB. Healthcare costs and workloss burden of patients with chemotherapy-associated peripheral neuropathy in breast, ovarian, head and neck, and nonsmall cell lung cancer. Chemother Res Pract. 2012;2012:913848. doi: 10.1155/2012/913848. Epub 2012 Mar 14. PMID 22482054
- [Background] Calhoun EA, Welshman EE, Chang CH, Lurain JR, Fishman DA, Hunt TL, Cella D. Psychometric evaluation of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (Fact/GOG-Ntx) questionnaire for patients receiving systemic chemotherapy. Int J Gynecol Cancer. 2003 Nov-Dec;13(6):741-8. doi: 10.1111/j.1525-1438.2003.13603.x. PMID 14675309